CLINICAL TRIAL: NCT03770247
Title: Direct Intraoperative Injection Versus Percutaneous CT Guided Celiac Plexus Neurolysis in Unresectable Pancreatic Cancer ; Randomized Controlled Study
Brief Title: Intraoperative Versus CT Guided Celiac Plexus Neurolysis in Unresectable Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MD ∕ 17.08.53
Record Dates: First submitted 2018-12-03; First posted 2018-12-10 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intraoperative group (IOCPN group) (Experimental): Intraoperative celiac plexus neurolysis Before closure of the abdomen the surgeon will expose the aorta at the level of the celiac trunk.With the stomach retracted inferiorly, the index and second finger of the surgeon's left hand straddle the aorta with the index finger placed on the splenic artery and the second finger on the common hepatic artery. we will use of a 20- gauge spinal needle (in contrast to the usual short intravenous needle) allows better visualization and access to this area, especially in deep patients, while a 10 ml syringe permits the surgeon to control the injection with the right hand alone.(10) Twenty ml of 90 % alcohol, five ml lidocaine 2%, five mg dexamethasone will be injected in each side of the aorta after aspiration to exclude intravascular or subarachnoid injection.
  Interventions: Procedure: Intraoperative celiac plexus neurolysis
- CT group (CTCPN group) (Active Comparator): CT guided celiac plexus neurolysis After one week of the operation and the patient completely awake, the patient will be transferred to CT lab. The procedure will be done after attachment of basic monitors and transfusion of 500 ml saline in 20 G cannula before starting the procedure and the patient will be given 5 mg midazolam as a sedation. The procedure will be done by anesthetist and radiologist who had a good experience in celiac plexus neurolysis. In our study we will use the classic posterior bilateral approach. The patient will be in the prone position. After sterilization of the back by chlorohixidine 10 % , subcutaneous injection of 5 ml lidocaine as a local anaesthesia until a wheel will be formed then the procedure will be done. We will use 20 G Chiba needle under guidance of CT. Twenty ml of 95% alcohol , five ml lidocaine 2 % and five mg dexamethasone in each side of the aorta after aspiaration to exclude intravascular injection and subarachnoid injection
  Interventions: Procedure: CT guided celiac plexus neurolysis

INTERVENTIONS:
Procedure: Intraoperative celiac plexus neurolysis — neurolysis of celiac plexus by intraoperative techniques
  Arms: intraoperative group (IOCPN group)
Procedure: CT guided celiac plexus neurolysis — Neurolysis of celiac plexus percutaneously by CT guidance
  Arms: CT group (CTCPN group)

SUMMARY:
Many studies had stated that the coeliac plexus neurolysis (CPN) is a safe and effective treatment method of pain associated with pancreatic cancer. The neurolytic injectate is usually alcohol 50-100%; however, phenol >5% is also possible to use. Nowadays, there are several techniques to access the coeliac plexus (per cutaneous using fluoroscopy or computed tomographic imaging (CT), surgical and endoscopic ultrasound). However, the percutaneous computed tomography guided technique is the gold standard technique, it has multiple drawbacks as availability and cost of imaging modality, exposure to radiation and multiple complications.Surgical technique in spite of being easy, cheap but there is a controversy about its efficacy. Also there is no head to head comparison between the surgical technique and the percutaneous technique.In this study we hypothesized that intraoperative technique has the same efficacy of percutaneous celiac block technique with less complication and cost

DETAILED DESCRIPTION:
This study aimed to compare the efficacy of the surgical technique versus the per cutaneous computed tomographic guided technique of celiac plexus neurolysis for pain management in unresectable pancreatic cancer . all patients suffering from pain of pancreatic cancer with VAS≥5 undergoing laparotomy and proved to be unresectable either undergoing biopsy or bypass surgery will receive celiac plexus neurolysis either intraoperative or post operative CT guided . All patients will be managed by systemic analgesic if the block not sufficient . In this study we will give the patient the analgesic according to WHO recommendation as starting by non steroidal anti inflammatory drugs as diclofenac sodium, if it is not sufficient we will give them opioids as tramadol, and for neuropathic pain gabapentin. All drugs will be given with escalating dose . Failed block defined as change in VAS between VAS BASELINE AND ONE MONTH ≤ 3 may need to repeat the block by percutaneous technique .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients suffering of pain from pancreatic cancer with baseline VAS≥5, scheduled for surgical assessment
* patients proven histololgically to be unresectable
* patients undergoing either biopsy or bypass surgery

Exclusion Criteria:

* patient with resectable tumour will be excluded.
* Patient with coagulopathy.
* patient with aortic aneurysm.
* patient with any disease contraindicating any sympathetic blockade as advanced cardiac disease .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
assesment of efficacy in pain palliation by change in VAS after one month | one month
  change in visual analogue scale ( VAS) after one month visual analogue scale is pain scale from 0 to 10 , 0 no pain , 10 maximum pain lower VAS better than higher .a positive responce defined as decrease of VAS of equal or more than 3

SECONDARY OUTCOMES:
incidence of complication | one month
  report the occurrence of complication as headache , diarrhea , vomiting , back pain
total analgesic consumption | 6 month
  the amount of analgesic required
duration of pain palliation | 6 month
  change of visual analogue scale from baseline for 6 months visual analogue scale represent pain from 0 no pain to 10 maximum pain
need of other injection | 6 months
  if failure of intervention occured patient may need another intervention

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M. Shams, MD, Study Director — : Professor of Anesthesia and Surgical Intensive Care; Mahmoud M. Elsedeiq, MSc, Principal Investigator — assistan lecturer of Anesthesia and Surgical Intensive Care; Mohamed A. Ghanim, MD, Study Chair — Assistant Professor of Anesthesia and Surgical Intensive Care; Ibrahim I. Abd El-basir, MD, Study Chair — Lecturer of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura university , gastrointestinal surgery center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided